CLINICAL TRIAL: NCT02860338
Title: Retrospective Analysis of the Comparative Effectiveness of MCI and Dementia Treatment Protocols in a Community-based Specialty Dementia Practice
Brief Title: COMPARATIVE EFFECTIVENESS OF MCI and DEMENTIA TREATMENTS IN A COMMUNITY-BASED DEMENTIA PRACTICE
Status: Completed | Type: Observational
Sponsor: Clionsky Neuro Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNS 2012-004
Record Dates: First submitted 2016-07-29; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Mild Cognitive Impairment; Dementia; Hypoxia; Hyperhomocysteinemia; Vitamin B 12 Deficiency; Iron Deficiency; Anemia; TBI; Neurodegenerative Disorders; Alzheimer's Disease; Vascular Dementia; Brain Injuries; Tauopathies; Parkinson's Disease; Lewy Body Dementia; Frontotemporal Dementia; TDP-43 Proteinopathies
Keywords: Psuedobulbar affect, PBA
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Hypoxia; Hyperhomocysteinemia; Vitamin B 12 Deficiency; Iron Deficiencies; Anemia; Neurodegenerative Diseases; Alzheimer Disease; Dementia, Vascular; Brain Injuries; Tauopathies; Parkinson Disease; Lewy Body Disease; Frontotemporal Dementia; TDP-43 Proteinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GROUP 1- CNS Protocol: Patients in a specialized dementia practice. Evaluated and treated for hypoxia, elevated BNP, hyperhomocysteinemia, B 12 deficiency as measured by elevated methymalonic acid, Vitamin D 25-OH deficiency, elevated CRP, and decreased IGF-1, and other metabolic abnormalities.
  Treated with maximal doses of acetylcholinesterase inhibitors, memantine, methylfolate/methylB12/N-acetylcysteine, dextromethorphan/quinidine, and SSRI's; dose and duration based on protocol.
- GROUP 2- Community Care: Patients referred to a neuropsychology practice for cognitive evaluation and treated for MCI or dementia by their primary care clinician or non-dementia specialist according to specific provider's usual practice pattern.

SUMMARY:
This retrospective study is a more extensive, confirmatory analysis of the cognitive and functional outcomes initially seen in 2 groups of MCI/dementia patients in Springfield, MA and compares specialized dementia care and a comprehensive treatment approach versus usual care delivered in a non-specialist setting.

The first group of patients (n= 328) was seen by a dementia specialist, who utilized a standardized assessment and treatment protocol (CNS). This included comprehensive identification and treatment of hypoxia, sleep-disorders, and other cognitively-impairing metabolic conditions as well as maximally- dosed FDA-approved medications for dementia, depression, and PBA.

The second group of patients (n= 280) was seen by non-dementia specialists in the community and received usual care which did not include comprehensive assessment or treatment of underlying metabolic derangements or maximal utilization of currently available medications.

This study, evaluating date from a larger cohort (n>800) of specialist-treated cognitively-impaired patients, will further examine the hypothesis that a comprehensive dementia treatment protocol yields cognitive stabilization and/or improvement using already available dementia drugs when compared with usual community care.

DETAILED DESCRIPTION:
From 2008-2013 more than 5,000 patients have been seen by a community-based internist/psychiatrist specializing in treating cognitively impaired adults suffering from MCI or dementia due to Alzheimer's Disease, vascular dementia, combined DAT/VAD, FTD, PD, LBD, as well as dementia due to traumatic brain injury (TBI), alcoholism and autoimmune diseases.

Cohort 1 includes patients from this specialist practice who were extensively evaluated with a standardized protocol assessment aimed at identifying all reversible and treatable conditions adversely affecting cognition, and achieving maximum diagnostic accuracy with respect to the underlying dementia pathology. The protocol included physical and mental status examinations, neuroimaging (PET scans and/or MRI's with volumetrics), lab tests, overnight pulse oximetry, in-lab and ambulatory polysomnography, and gold standard neuropsychological testing as well as rapid, in-office cognitive testing. The comprehensive treatment protocol attempted correction of all modifiable and metabolic derangements, and utilized maximally tolerated FDA approved medications and devices.

Cohort 2 includes patients who were referred by their primary care clinicians or other non-dementia specialists to a neuropsychology practice for a standardized cognitive evaluation as part of usual care, but were not treated by a dementia specialist.

This in-depth retrospective analysis is the first attempt to evaluate the comparative effectiveness of dementia drugs and other treatment interventions in a cognitively impaired patient group whose baseline metabolic abnormalities were identified, treated and maintained optimally throughout the course of care versus a patient group not so intensively assessed or managed.

Outcome measures include objective cognitive testing and functional and behavioral assessments correlated with prescribed standard dementia medications, reductions in benzodiazepine, narcotic and antipsychotic use, as well as with baseline and interval measures of oxygenation adequacy, BNP, CRP, IGF-1, homocysteine, methylmalonic acid, iron status, Vitamin D 25-OH, and utilization of oxygen and positive airway pressure treatment.

ELIGIBILITY:
Inclusion Criteria:

* individuals presenting for assessment and treatment of cognitive impairment, either by self-identification, report by family or caregivers, or upon referral from another physician.

Exclusion Criteria:

* individuals who were not fluent in English and for whom a translator was not available.
* individuals who were blind

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Consecutive patients presenting for care for cognitive impairment in a non-academic, non-hospital based, dementia specialty practice in Springfield, MA Cohort 2: Convenience sample of patients referred to neuropsychological testing and treated by non-dementia specialists in Springfield, MA
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cognitive testing - Memory Orientation Screening Test (MOST) | At each office visit, for 96 months, until patient left the practice, or until date of death

SECONDARY OUTCOMES:
Resting and ambulatory pulse oximetry in office | At each office visit, for 96 months, until patient left the practice, or until date of death
  Recording of the pulse oximetry data from a standard Nonan pulse oximeter while the patient is at rest and/or ambulation at office visits made by the patient as determined by usual patient care in a naturalistic setting
Nocturnal pulse oximetry | Ordered and Initial office visit or subsequent patient visits, for 96 months, until the patient left the practice, or until the date of death.
  Recording of SpO2, baseline, nadir, time <=88%, oxygen desaturation index, heart rate range, nadir heart rate, maximum heart rate using standardized, FDA-device approved, commercially available nocturnal pulse oximeters
Polysomnography in-lab and ambulatory ( in patient's residence) | Initial study ordered at first or subsequent office visit for for 96 months, until the patient left the practice, or until the date of death.
  Polysomnography date obtained from standardized, commercially available, FDA approved instruments, including: number of nights studied (1-3), apnea-hypoxia index (AHI), nadir heart rate, heart rate range, nadir SpO2, diagnosis reported
Laboratory values: Chem 20, CBC/diff, BNP, CRP, iron, iron/TIBC, ferritin, homocysteine, methylmalonic acid, Vitamin D 25-OH, RPR/FTA-ABS/TPPA, IGF-1 | Ordered at initial and subsequent office visits for 96 months, until patient left the practice, or until date of death

OTHER OUTCOMES:
Medications - prescribed | Ordered ar Initial office visit and any subsequent visits for Ordered at initial and subsequent office visits for 96 months, until patient left the practice, or until date of death
  Initiation, duration of use, dosing levels, adverse side effects, discontinuation/reason for discontinuation of prescribed dementia medications or other drugs, including but not limited to donepezil, rivastigmine, galantamine, memantine, methlyfolate/methylB12/N-acetylcysteine, cholecalciferol, dextromethorphan/quinidine, eszopiclone, citalopram, escitalopram, and sertraline
Oxygen - prescribed | Ordered at either at initial or subsequent office visit for a period of 96 months, or until patient left the practice, or until date of death
  Initiation, duration, and reason for discontinuation of O 2 nasal cannula supplementation either 24 x 7, or only while sleeping
Diagnosis: Obstructive/Central/Complex Sleep Apnea CPAP- Continuous Positive Airway Pressure or Bi-PAP | CPAP ordered at either at initial or subsequent office visit for a period of 96 months, or until patient left the practice, or until date of death
  Initiation, method of accustomization/desensitzation, duration of use, compliance, and reason for discontinuation
Diagnosis: Bradycardia/tachycardia | Recorded at all office visits or overnight testing for a period of 96 months, or until patient left the practice, or until date of death
  Heart rate under 60 or over 100 Correlation with rate control medications and acetylcholinesterase inhibitor
Discontinuation of cognitively impairing medications or other high risk medications (Beers criteria): benzodiazepines, narcotics, anticholinergics, and antipsychotics | At initial office visit and all subsequent visits for a period of 96 months, or until patient left the practice, or until date of death
  Class of drug, dose, date of discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Emily F Clionsky, M.D., Principal Investigator — Clionsky Neuro Systems Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clionsky MI, Clionsky E. Development and validation of the Memory Orientation Screening Test (MOST): A better screening test for dementia. Am J Alzheimers Dis Other Demen. 2010 Dec;25(8):650-6. doi: 10.1177/1533317510386216. PMID 21131671
- [Background] The Memory Orientation Screening Test accurately separates Normal from MCI and Demented Elder in a prevalence-stratified sample. Journal of Alzheimer's Disease and Parkinsonism. 2013 vol 3(1). http://dx.doi,org/10.4172/2161-04601000109
- [Background] Clionsky M, Clionsky E. Psychometric equivalence of a paper-based and computerized (iPad) version of the Memory Orientation Screening Test (MOST(R)). Clin Neuropsychol. 2014;28(5):747-55. doi: 10.1080/13854046.2014.913686. Epub 2014 May 12. PMID 24815733
- See also: AAN 2014 moderator -presented poster — https://www.researchgate.net/publication/264557391_Comparative_Effectiveness_of_an_Advanced_Treatment_Protocol_for_Dementia_vs_Standard_Community_Care